CLINICAL TRIAL: NCT03681951
Title: A Phase I/II, Open-Label Study to Investigate the Safety, Clinical Activity, Pharmacokinetics, and Pharmacodynamics of GSK3145095 Administered Alone and in Combination With Anticancer Agents Including Pembrolizumab in Adult Participants With Selected Advanced Solid Tumors
Brief Title: First-time-in-human (FTIH) Study of GSK3145095 Alone and in Combination With Other Anticancer Agents in Adults With Advanced Solid Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated following an internal review of the company's current research and development portfolio.
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 205013
Record Dates: First submitted 2018-09-10; First posted 2018-09-24 (Actual); Results first posted 2020-07-31 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Neoplasms, Pancreatic
Keywords: Anticancer Agents; FTIH; Pembrolizumab; Rip1K; GSK3145095; Dose Escalation; Immunotherapy resistance; Dose Expansion; RECIST 1.1; Advanced solid tumors; Innate immunity
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Part 1 dose escalation will administer escalating doses of GSK3145095 as monotherapy only. Part 2 will combine escalating doses of GSK3145095 with 200 mg pembrolizumab. Dose escalation of GSK3145095 will begin at least one level below the highest dose shown to have an acceptable toxicity profile in at least 3 subjects in Part 1. Part 3 will enroll subjects treated with one or more dose levels of GSK3145095 in combination with 200 mg pembrolizumab. Part 4 will investigate the combination of additional anticancer agents with one or more doses of GSK3145095 identified as safe in Part 1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: Dose Escalation - GSK3145095 monotherapy (Experimental): In Part 1, advanced or metastatic PDAC will be enrolled. Part 1 will be using escalating doses of GSK3145095 (total daily dose of 100 mg, 200 mg, 400 mg, 800 mg, and 1600 mg) orally as monotherapy for up to 2 years. For each dose level, subjects will receive a single dose of half the total daily dose on Day 1; and as BID (total daily dose divided in two equal doses) starting from Day 2.
  Interventions: Drug: GSK3145095
- Part 2: Dose Escalation - GSK3145095 + pembrolizumab (Experimental): In Part 2, subjects with selected solid tumors, including but not limited to, PDAC, NSCLC, TNBC and/or melanoma will be enrolled. Part 2 will be using GSK3145095 combination escalation to start at least one dose level below the highest dose of GSK3145095 shown to be safe in Part 1, orally BID for up to 2 years along with pembrolizumab 200 mg intravenous (IV) every 3 weeks (Q3W) for up to 2 years.
  Interventions: Drug: GSK3145095; Drug: Pembrolizumab
- Part 3: Dose Expansion - GSK3145095 + pembrolizumab (Experimental): In Part 3, subjects with selected solid tumors will be enrolled. Part 3 will be using GSK3145095 at one or two dose levels shown to be tolerable in Part 2 orally BID for up to 2 years along with pembrolizumab 200 mg IV Q3W for up to 2 years.
  Interventions: Drug: GSK3145095; Drug: Pembrolizumab
- Part 4: Dose Expansion - GSK3145095 + anticancer agent (Experimental): In Part 4, subjects with selected solid tumors will be enrolled. Part 4 will be using GSK3145095 at one or two dose levels shown to be tolerable in Part 2 orally BID for up to 2 years along with combination of additional anticancer agents.
  Interventions: Drug: GSK3145095

INTERVENTIONS:
Drug: GSK3145095 — GSK3145095 will be available as capsule (size 1 containing 5 to 25 mg GSK3145095 and size 0 containing 25 to 75 mg GSK3145095) or tablet (25, 50, 200 mg white to slightly covered round/oval shaped coated) for oral administration in the fasted stated with approximately 200 milliliters (mL) of water.
Drug: Pembrolizumab — Pembrolizumab will be available as solution for infusion (100 milligrams/ 4 milliliter) at a dose of 200 mg via IV infusion for 30 minutes (given the variability of infusion pumps from site to site, a window of -5 minutes and +10 minutes is permitted i.e., infusion time is 25 to 40 minutes).
  Arms: Part 2: Dose Escalation - GSK3145095 + pembrolizumab; Part 3: Dose Expansion - GSK3145095 + pembrolizumab

SUMMARY:
In an unbiased CRISPR screen, RIPK1 was identified as a top gene contributing to immunotherapy resistance. In addition, RIPK1 has been reported to drive pancreatic oncogenesis. In murine models, inhibition of RIPK1 kinase activity in the pancreatic tumor microenvironment leads to the replacement of tumor-permissive myeloid infiltrates with innate cells that promote an effective antitumor response by adaptive cells. The investigators hypothesize that inhibition of RIPK1 in human pancreatic cancer subjects will modulate the immune infiltrate to sensitize tumors to checkpoint blockade.

DETAILED DESCRIPTION:
Study 205013 is a Phase 1 FTIH study of GSK3145095 alone and in combination with other anticancer agents including pembrolizumab in subjects with pancreatic ductal adenocarcinoma (PDAC) and other selected tumors. The study includes up to 4 parts: Part 1 dose escalation will be conducted in approximately 30 adult subjects with advanced or metastatic PDAC using escalating doses of GSK3145095 as monotherapy only. Part 2 will combine escalating doses of GSK3145095 with 200 milligram (mg) pembrolizumab. Dose escalation of GSK3145095 will begin at least one level below the highest dose shown to have an acceptable toxicity profile in at least 3 subjects in Part 1. Part 2 may be conducted in a broader population of selected solid tumors using a combination of escalating doses of GSK3145095 and 200 mg pembrolizumab. Part 3 will enroll subjects treated with one or more dose levels of GSK3145095 in combination with 200 mg pembrolizumab. Part 4 will investigate the combination of additional anticancer agents with one or more doses of GSK3145095 identified as safe in Part 1. Up to approximately 220 subjects will be treated in the study. Parts 1 and 2 will each treat up to approximately 30 subjects. Parts 3 and 4 will treat up to approximately 160 subjects (up to 80 subjects in each Part). The total duration of the study is expected to last up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must provide signed, written informed consent.
* Male and female subjects, age >=18 years (at the time consent is obtained). a) Male subjects are eligible to participate if they agree to the following during the study treatment period and for at least 15 days (Part 1) and 120 days (Parts 2-4) after the last dose of study treatment: Refrain from donating sperm, be abstinent from heterosexual or homosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent or must agree to use contraception/barrier: male condom and female partner to use an additional highly effective contraceptive method with a failure rate of <1 percent per year. b) female subjects are eligible to participate if they are not either pregnant or breastfeeding, and at least one of the following conditions applies: is not a woman of childbearing potential (WOCBP), is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1 percent per year), with low user dependency during the study treatment period and for at least 15 days (Part 1) and 120 days (Parts 2-4) after the last dose of study treatment and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during this period. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study treatment. Hormonal contraception may be susceptible to interaction with the study drug, which may reduce the efficacy of the contraceptive method. Therefore, a barrier method is also required for subjects using a hormonal option (including hormonal intrauterine device [IUD], oral contraceptive pills/ patch/ vaginal inserts, and hormonal implants) and both highly effective methods of contraception should be utilized during the treatment period and for at least 15 days (Part 1) and 120 days (Parts 2-4) after the last dose of study treatment.If a highly effective non-hormonal method is used, then only one method of contraception is required (by a female participant or partner of a male participant; in either situation the male partner must still use a male condom in addition) during the treatment period and for at least 15 days (Part 1) and 120 days (Parts 2-4) after the last dose of study treatment. A WOCBP must have a negative highly sensitive pregnancy test (urine or serum) as required by local regulations) within 24 hours before the first dose of study intervention. If a urine test cannot be confirmed as negative (e.g., an ambiguous result), a serum pregnancy test is required. In such cases, the subject must be excluded from participation if the serum pregnancy result is positive. If the subject hasn't been on an acceptable method of contraception for at least 2 weeks prior to start of therapy, pregnancy testing must be done weekly for the first month of treatment. Additional requirements for pregnancy testing during and after study treatment. The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
* Histological documentation of locally advanced, recurrent or PDAC (Part 1), non-small cell lung cancer (NSCLC), triple negative breast cancer (TNBC), or melanoma (Part 2) that has progressed after standard therapy appropriate for the specific tumor type, or for which standard therapy has proven to be ineffective, intolerable, or is considered inappropriate. Subjects should have received at least one, but not more than 2 prior lines of therapy for advanced disease including both standards of care and investigational therapies. Subjects whose cancers harbor molecular alterations for which targeted therapy is standard of care should have received health authority-approved appropriate targeted therapy for their tumor types before enrollment.
* All subjects in Parts 1 and 2 must consent to provide a fresh biopsy during screening of a primary tumor lesion or from other metastases (e.g. liver, lung, etc.), and a second biopsy after approximately 5 weeks of treatment.
* Measurable disease per RECIST version 1.1. Palpable lesions that are not measurable by radiologic or photographic evaluations may not be utilized as the only measurable lesion. Subjects are encouraged to provide a pre-Baseline scan (within 24 weeks before the Baseline scan) to support exploratory investigation of tumor growth kinetics.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 to 1.
* Life expectancy of at least 12 weeks.
* Adequate organ function.
* QT duration corrected for heart rate by Fridericia's formula (QTcF) <450 milliseconds (or QTcF <480 milliseconds for subjects with bundle branch block).

Exclusion Criteria:

* Prior treatment with the following agents: Agents affecting tumor associated macrophage function or number, including but not limited to inhibitors of Receptor-interacting protein 1 (RIP1), Receptor-interacting protein 3 (RIP3), Colony stimulating factor 1 receptor (CSFR-1), C-C chemokine receptor type 2 (CCR2), and Cluster of differentiation 40 (CD40). Other anticancer therapy, including chemotherapy, targeted therapy, and biological therapy, within 14 days or 5 half-lives (from last dose of prior treatment to first dose of GSK3145095), whichever is shorter. Prior radiation therapy is permissible if at least one non-irradiated measurable lesion is available for assessment via RECIST version 1.1. No washout after palliative radiation is required. Investigational therapy within 14 days or 5 half-lives (from last dose of prior treatment to first dose of GSK3145095), whichever is shorter.
* Prior allogeneic or autologous bone marrow transplantation or other solid organ transplantation.
* Toxicity from previous treatment: Subjects whose toxicity related to prior treatment has not resolved to <=Grade 1 (except alopecia, hearing loss, Grade <=2 neuropathy or endocrinopathy managed with replacement therapy) are not eligible.
* Malignancy other than disease under study, except as noted: Subject with any other malignancy from which the subject has been disease-free for more than 2 years and, in the opinion of the principal investigators and GlaxoSmithKline (GSK) Medical Monitor, will not affect the evaluation of the effects of this clinical trial treatment on currently targeted malignancy, can be included in this clinical trial.
* Major surgery <=4 weeks before the first dose of study treatment. Subjects must have also fully recovered from any surgery (major or minor) and/or its complications before initiating study treatment.
* Active autoimmune disease that has required systemic treatment within the last 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Concurrent medical condition requiring the use of systemic immunosuppressive medications within 28 days before the first dose of study treatment. Physiologic doses of corticosteroids for treatment of endocrinopathies or steroids with minimal systemic absorption, including topical, inhaled, or intranasal corticosteroids, may be continued if the subject is on a stable dose.
* Active infection (including active herpes zoster infection), known human immunodeficiency virus infection, or positive test for hepatitis B surface antigen or hepatitis C.
* Current active liver or biliary disease (except for Gilbert's syndrome or asymptomatic gallstones, liver metastases, or otherwise stable chronic liver disease per investigator assessment).
* Known current drug or alcohol abuse.
* Recent history (within the past 6 months) of acute diverticulitis, inflammatory bowel disease, intra-abdominal abscess, or gastrointestinal obstruction.
* Receipt of any live vaccine within 4 weeks before starting study treatment.
* Recent history of allergen desensitization therapy within 4 weeks before starting study treatment (applies to subjects enrolled in Parts 2 and 3 only).
* History or evidence of cardiovascular risk including any of the following: recent (within the past 6 months) history of serious uncontrolled cardiac arrhythmia or clinically significant electrocardiogram (ECG) abnormalities including second degree (Type II) or third degree atrioventricular block. Documented cardiomyopathy, myocardial infarction, acute coronary syndromes (including unstable angina pectoris), coronary angioplasty, stenting, or bypass grafting within the past 6 months before beginning screening. Documented congestive heart failure (Class II, III, or IV) as defined by the New York Heart Association functional classification system. Recent (within the past 6 months) history of symptomatic pericarditis.
* Current or history of idiopathic pulmonary fibrosis, interstitial lung disease, or organizing pneumonia.
* History of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Recent history (within 14 days) of ascites or pleural effusions requiring drainage.
* Any serious and/or unstable pre-existing medical, psychiatric disorder, or other condition that could interfere with the subjects safety, obtaining informed consent, or compliance to the study procedures.
* Is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling or child) who is investigational site or sponsor staff directly involved with this trial, unless prospective Institutional Review Board (IRB) approval (by chair or designee) is given allowing exception to this criterion for a specific subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2019-08-13 (Actual); Study Completion 2019-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- United States (4):
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label study to investigate the safety, clinical activity, pharmacokinetics, and pharmacodynamics of GSK3145095 administered alone and in combination with anticancer agents including Pembrolizumab in adult participants with selected advanced solid tumors.
Pre-assignment Details: Total 8 participants were included in part 1 of the study across United States. This study was terminated during Part 1 (Monotherapy dose escalation [DE]) and hence Part 2,3,4 were not conducted following an internal review of the company's current research and development portfolio.
Groups:
- Part 1-GSK3145095 50 mg BID: Participants received a single 50 milligram (mg) dose of GSK3145095 orally on Day 1. From study day 2, participants then received total daily dose of 100 mg GSK3145095 orally given as 50 mg twice a day (BID).
- Part 1-GSK3145095 100 mg BID: Participants were to receive a single 100 mg dose of GSK3145095 orally on Day 1. From study Day 2, participants were to receive 200 mg GSK3145095 given as 100 mg BID.
- Part 1-GSK3145095 200 mg BID: Participants were to receive a single 200 mg dose of GSK3145095 orally on Day 1. From study Day 2, participants were to receive 400 mg GSK3145095 given as 200 mg BID.
- Part 1-GSK3145095 400 mg BID: Participants were to receive a single 400 mg dose of GSK3145095 orally on Day 1. From study Day 2, participants were to receive 800 mg dose of GSK3145095 given as 400 mg BID
- Part 1-GSK3145095 800 mg BID: Participants were to receive a single 800 mg dose of GSK3145095 orally on Day 1. From study Day 2, participants were to receive 1600 mg dose of GSK3145095 given as 800 mg BID.
- Part 2- GSK3145095+ Pembrolizumab 200 mg: Part 2 was to be initiated after evaluation of safety and toxicity data of Part 1. Participants in this combination therapy arm were planned to receive GSK3145095 at one dose level below the highest dose shown to have an acceptable toxicity profile in at least 3 participants in Part 1 in combination with 200 mg pembrolizumab as Intravenous (IV) infusion over 30 minutes (min) for every 3 weeks.
- Part 3- GSK3145095+ Pembrolizumab 200 mg: Part 3 was to be initiated after evaluation of safety and toxicity data of part 2. Participants in this combination therapy arm were planned to receive GSK3145095 at recommended dose level determined during Part 2, with 200 mg pembrolizumab as IV infusion for every 3 weeks
- Part 4- GSK3145095+ Anticancer Agent: In Part 4, participants were planned to receive GSK3145095 at recommended dose level determined during Part 2, in combination with anticancer agent.
Period: Part1: Monotherapy DE (Up to Day 95)
Arm/Group | Part 1-GSK3145095 50 mg BID | Part 1-GSK3145095 100 mg BID | Part 1-GSK3145095 200 mg BID | Part 1-GSK3145095 400 mg BID | Part 1-GSK3145095 800 mg BID | Part 2- GSK3145095+ Pembrolizumab 200 mg | Part 3- GSK3145095+ Pembrolizumab 200 mg | Part 4- GSK3145095+ Anticancer Agent
Started | 8 | 0 (No participant was enrolled in this arm as study was terminated during cohort "GSK3145095 50mg BID") | 0 (No participant was enrolled in this arm as study was terminated during cohort "GSK3145095 50mg BID".) | 0 (No participant was enrolled in this arm as study was terminated during cohort "GSK3145095 50mg BID") | 0 (No participant was enrolled in this arm as study was terminated during cohort "GSK3145095 50mg BID") | 0 (Part 2 was not initiated as this study was terminated during Part 1) | 0 (Part 3 was not initiated as this study was terminated during Part 1) | 0 (Part 4 was not initiated as this study was terminated during Part 1)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part2:Combination Therapy(Upto 2yr90day)
Arm/Group | Part 1-GSK3145095 50 mg BID | Part 1-GSK3145095 100 mg BID | Part 1-GSK3145095 200 mg BID | Part 1-GSK3145095 400 mg BID | Part 1-GSK3145095 800 mg BID | Part 2- GSK3145095+ Pembrolizumab 200 mg | Part 3- GSK3145095+ Pembrolizumab 200 mg | Part 4- GSK3145095+ Anticancer Agent
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3:Dose Expansion (Up to 2yr90day)
Arm/Group | Part 1-GSK3145095 50 mg BID | Part 1-GSK3145095 100 mg BID | Part 1-GSK3145095 200 mg BID | Part 1-GSK3145095 400 mg BID | Part 1-GSK3145095 800 mg BID | Part 2- GSK3145095+ Pembrolizumab 200 mg | Part 3- GSK3145095+ Pembrolizumab 200 mg | Part 4- GSK3145095+ Anticancer Agent
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 4: Dose Expansion(Up to 2 yr90day)
Arm/Group | Part 1-GSK3145095 50 mg BID | Part 1-GSK3145095 100 mg BID | Part 1-GSK3145095 200 mg BID | Part 1-GSK3145095 400 mg BID | Part 1-GSK3145095 800 mg BID | Part 2- GSK3145095+ Pembrolizumab 200 mg | Part 3- GSK3145095+ Pembrolizumab 200 mg | Part 4- GSK3145095+ Anticancer Agent
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Part 1-GSK3145095 50 mg BID data is presented as study was terminated during Part 1 and hence Part 2, 3 and 4 were not initiated.
Groups:
- Part 3- GSK3145095+ Pembrolizumab 200mg: Part 3 was to be initiated after evaluation of safety and toxicity data of part 2. Participants in this combination therapy arm were planned to receive GSK3145095 at recommended dose level determined during Part 2, with 200 mg pembrolizumab as IV infusion for every 3 weeks.
- Total: Total of all reporting groups
Arm/Group | Part 1-GSK3145095 50 mg BID | Part 1-GSK3145095 100 mg BID | Part 1-GSK3145095 200 mg BID | Part 1-GSK3145095 400 mg BID | Part 1-GSK3145095 800 mg BID | Part 2- GSK3145095+ Pembrolizumab 200 mg | Part 3- GSK3145095+ Pembrolizumab 200mg | Part 4- GSK3145095+ Anticancer Agent | Total
Number analyzed (Participants) | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.5 (5.68) |  |  |  |  |  |  |  | 66.5 (5.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 |  |  |  |  |  |  |  | 4
  Male | 4 |  |  |  |  |  |  |  | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: BLACK OR AFRICAN AMERICAN | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Race: WHITE/CAUCASIAN/EUROPEAN HERITAGE | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  Race: MISSING | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Non-serious Adverse Events (AEs) and Serious Adverse Events (SAEs)-Part 1
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. SAE is defined as any untoward medical occurrence that, at any dose which results in death, is life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or other situations.
Time Frame: Up to Day 95
Population: All treated Population consisted of all participants who received at least one dose of GSK3145095. Study was terminated in Part-1 during first escalation cohort "GSK3145095 50 mg BID", hence subsequent escalation cohorts were not initiated.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1-GSK3145095 50 mg BID | Part 1-GSK3145095 100 mg BID | Part 1-GSK3145095 200 mg BID | Part 1-GSK3145095 400 mg BID | Part 1-GSK3145095 800 mg BID
Number analyzed (Participants) | 8 | 0 | 0 | 0 | 0
Participants
  Non-serious AEs | 8 |  |  |  |
  SAEs | 4 |  |  |  |

2. Primary Outcome: Number of Participants With Non-serious AEs and SAEs-Part 2
Description: as for outcome 1
Time Frame: Up to 2 years and 90 days
Population: All treated Population: Data were not collected for this endpoint as study was terminated during Part 1. Subsequent Part 2 was not initiated.
Groups:
- Part 2-GSK3145095+ Pembrolizumab 200 mg: Part 2 was to be initiated after evaluation of safety and toxicity data of Part 1. Participants in this combination therapy arm were planned to receive GSK3145095 at one dose level below the highest dose shown to have an acceptable toxicity profile in at least 3 participants in Part 1 in combination with 200 mg pembrolizumab as IV infusion over 30 minutes for every 3 weeks.
Arm/Group | Part 2-GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

3. Primary Outcome: Number of Participants With AEs by Severity Grades-Part 1
Description: All adverse events were analyzed using National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0. Graded from Grade 1: mild asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated, Grade 2: Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL), Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL, Grade 4: Life-threatening consequences; urgent intervention indicated, Grade 5: death related AE. Higher grade indicates more severe condition. Number of participants with maximum severity grades were presented.
Time Frame: Up to Day 95
Population: All treated Population: Study was terminated in Part-1 during first escalation cohort "GSK3145095 50 mg BID", hence subsequent escalation cohorts were not initiated.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1-GSK3145095 50 mg BID | Part 1-GSK3145095 100 mg BID | Part 1-GSK3145095 200 mg BID | Part 1-GSK3145095 400 mg BID | Part 1-GSK3145095 800 mg BID
Number analyzed (Participants) | 8 | 0 | 0 | 0 | 0
Participants
  Grade 1 | 0 |  |  |  |
  Grade 2 | 3 |  |  |  |
  Grade 3 | 4 |  |  |  |
  Grade 4 | 1 |  |  |  |
  Grade 5 | 0 |  |  |  |

4. Primary Outcome: Number of Participants With AEs by Severity Grades-Part 2
Description: All adverse events were to be analyzed using NCI-CTCAE Version 5.0. Graded from Grade 1: mild asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated, Grade 2: Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL, Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL, Grade 4: Life-threatening consequences; urgent intervention indicated, Grade 5: death related AE. Higher grade indicates more severe condition.
Time Frame: Up to 2 years and 90 days
Population: as for outcome 2
Arm/Group | Part 2-GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

5. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs)-Part 1
Description: All toxicities were graded using NCI-CTCAE version 5.0. An AE was considered a DLT if it occurred during the first 28 days of treatment, was considered by the investigator to be clinically relevant, and met one of the following DLT criteria: hematologic toxicity: Grade 4 neutropenia, febrile neutropenia, Grade 4 anemia, Grade 3 thrombocytopenia, Grade 3 thrombocytopenia with bleeding; Grade 3 or greater non-hematologic toxicity, any Grade 2 ocular toxicity requiring systemic steroids.
Time Frame: Up to Day 28
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1-GSK3145095 50 mg BID | Part 1-GSK3145095 100 mg BID | Part 1-GSK3145095 200 mg BID | Part 1-GSK3145095 400 mg BID | Part 1-GSK3145095 800 mg BID
Number analyzed (Participants) | 8 | 0 | 0 | 0 | 0
Participants | 0 |  |  |  |

6. Primary Outcome: Number of Participants With DLTs-Part 2
Description: as for outcome 5
Time Frame: Up to 28 days
Population: as for outcome 2
Arm/Group | Part 2-GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

7. Primary Outcome: Percentage of Participants Achieving Complete Response (CR) or Partial Response (PR) Based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 Criteria-Part 3
Description: A participant's disease status and determination of disease progression at post Baseline visits was to be evaluated by the local investigator's assessments by RECIST version 1.1. The overall response rate (ORR)-CR and PR was to be determined by the investigator assessment of the participants computed tomography (CT) or magnetic resonance imaging (MRI) using RECIST version 1.1 criteria for target lesions. ORR is defined as the percentage of participants with a best overall confirmed CR or PR at any time as per disease-specific criteria. PR is when there is at least 30 percent decrease in sum of the longest diameter of the target lesions. Complete Response is when there is disappearance of all non-nodal target lesions, with the short axes of any target lymph nodes reduced to <10 millimeters (mm).
Time Frame: Until response, disease progression, initiation of another anticancer therapy or death whichever is earlier (maximum follow-up up to 2 years 90 days)
Population: All treated Population: Data were not collected for this endpoint as study was terminated during Part 1. Subsequent Part 3 was not initiated.
Groups:
- Part 3 GSK3145095+ Pembrolizumab 200 mg: Part 3 was to be initiated after evaluation of safety and toxicity data of part 2. Participants in this combination therapy arm were planned to receive GSK3145095 at recommended dose level determined during Part 2, with 200 mg pembrolizumab as IV infusion for every 3 weeks.
Arm/Group | Part 3 GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

8. Primary Outcome: Percentage of Participants Achieving Complete Response or Partial Response Based on RECIST 1.1 Criteria-Part 4
Description: A participant's disease status and determination of disease progression at post Baseline visits was to be evaluated by the local investigator's assessments by RECIST version 1.1. The overall response rate (complete response and partial response) was to be determined by the investigator assessment of the participants CT or MRI using RECIST version 1.1 criteria for target lesions. ORR is defined as the percentage of participants with a best overall confirmed CR or PR at any time as per disease-specific criteria. Partial Response is when there is at least 30 percent decrease in sum of the longest diameter of the target lesions. Complete Response is when there is disappearance of all non-nodal target lesions, with the short axes of any target lymph nodes reduced to <10 mm.
Time Frame: Until response, disease progression, initiation of another anticancer therapy or death whichever is earlier (maximum follow-up up to 2 years and 90 days)
Population: All treated Population: Data were not collected for this endpoint as study was terminated during Part 1. Subsequent Part 4 was not initiated.
Groups:
- Part 4 GSK3145095+ Anticancer Agent: In Part 4, participants were planned to receive GSK3145095 at recommended dose level determined during Part 2, in combination with anticancer agent.
Arm/Group | Part 4 GSK3145095+ Anticancer Agent
Number analyzed (Participants) | 0

9. Secondary Outcome: Best Overall Response (BOR) Rate-Part 1
Description: Best overall response is defined as the best unconfirmed response (Complete Response [CR] > Partial Response [PR] > Stable Disease [SD] [or non-CR/non-PD] > Progressive Disease [PD] > Not Evaluable [NE]) from treatment start date until disease progression or initiation of new anti-cancer therapy, whichever is earlier, as assessed by the investigator per RECIST version 1.1 Criteria. The BOR rate is defined as the percentage of participants with each best unconfirmed response category. Participants with unknown or missing responses were treated as non-responders, i.e., these participants were included in the denominator when calculating percentages of response.
Time Frame: Until response, disease progression, initiation of another anticancer therapy or death whichever is earlier (maximum follow-up up to 95 days)
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1-GSK3145095 50 mg BID | Part 1-GSK3145095 100 mg BID | Part 1-GSK3145095 200 mg BID | Part 1-GSK3145095 400 mg BID | Part 1-GSK3145095 800 mg BID
Number analyzed (Participants) | 8 | 0 | 0 | 0 | 0
Percentage of participants
  Complete response | 0 |  |  |  |
  Partial response | 0 |  |  |  |
  Stable disease | 0 |  |  |  |
  Progressive disease | 62.5 |  |  |  |
  Not evaluable | 37.5 |  |  |  |

10. Secondary Outcome: Best Overall Response (BOR) Rate-Part 2
Description: Best overall response is defined as the best unconfirmed response (CR > PR > SD [or non-CR/non-PD] > PD] > NE) from treatment start date until disease progression or initiation of new anti-cancer therapy, whichever is earlier, as assessed by the investigator per RECIST 1.1 Criteria. The BOR rate is defined as the percentage of participants with each best unconfirmed response category. Participants with unknown or missing responses were treated as non-responders, i.e., these participants were included in the denominator when calculating percentages of response.
Time Frame: as for outcome 8
Population: as for outcome 2
Arm/Group | Part 2-GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

11. Secondary Outcome: Progression-free Survival (PFS)-Part 3
Description: PFS is defined as time from the date of first dose to the date of disease progression according to clinical or radiological assessment or death due to any causes, whichever occurs earliest. If the participant received subsequent anti-cancer therapy prior to the date of documented events, PFS was to be censored at the last adequate assessment (e.g., assessment where visit level response is confirmed response, partial response or stable disease) prior to the initiation of therapy. Otherwise, if the participant did not have a documented date of event, PFS was to be censored at the date of the last adequate assessment.
Time Frame: Until disease progression or death whichever is earlier (maximum follow-up up to 2 years and 90 days)
Population: as for outcome 7
Arm/Group | Part 3 GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

12. Secondary Outcome: Progression-Free Survival (PFS) -Part 4
Description: as for outcome 11
Time Frame: Until disease progression or death whichever is earlier (maximum follow-up up to 2 years and 90 days)
Population: as for outcome 8
Arm/Group | Part 4 GSK3145095+ Anticancer Agent
Number analyzed (Participants) | 0

13. Secondary Outcome: Overall Survival -Part 3
Description: Overall survival is defined as time from the date of first dose to the date of death due to any cause. If a participant does not have a documented date of death, time of death is censored at the date of last contact.
Time Frame: Until death (maximum follow-up up to 2 years and 90 days)
Population: as for outcome 7
Arm/Group | Part 3 GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

14. Secondary Outcome: Overall Survival -Part 4
Description: as for outcome 13
Time Frame: Until death (maximum follow-up up to 2 years and 90 days)
Population: as for outcome 8
Groups:
- Part 4 GSK3145095 200 mg + Anticancer Agent: In Part 4, participants were planned to receive GSK3145095 at recommended dose level determined during Part 2, in combination with anticancer agent.
Arm/Group | Part 4 GSK3145095 200 mg + Anticancer Agent
Number analyzed (Participants) | 0

15. Secondary Outcome: Number of Participants With Non-serious AEs and SAEs-Part 3
Description: as for outcome 1
Time Frame: Up to 2 years and 90 days
Population: as for outcome 7
Arm/Group | Part 3 GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

16. Secondary Outcome: Number of Participants With Non-serious AEs and SAEs-Part 4
Description: as for outcome 1
Time Frame: Up to 2 years and 90 days
Population: as for outcome 8
Groups:
- Part 4 GSK3145095 + Anticancer Agent: In Part 4, participants were planned to receive GSK3145095 at recommended dose level determined during Part 2, in combination with anticancer agent.
Arm/Group | Part 4 GSK3145095 + Anticancer Agent
Number analyzed (Participants) | 0

17. Secondary Outcome: Number of Participants With AEs by Severity Grades-Part 3
Description: All adverse events were planned to be analyzed using NCI-CTCAE Version 5.0. Graded from Grade 1: mild asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated, Grade 2: Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL, Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL, Grade 4: Life-threatening consequences; urgent intervention indicated, Grade 5: death related AE. Higher grade indicates more severe condition.
Time Frame: Up to 2 years and 90 days
Population: as for outcome 7
Arm/Group | Part 3 GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

18. Secondary Outcome: Number of Participants With AEs by Severity Grades-Part 4
Description: as for outcome 17
Time Frame: Up to 2 years and 90 days
Population: as for outcome 8
Arm/Group | Part 4 GSK3145095 + Anticancer Agent
Number analyzed (Participants) | 0

19. Secondary Outcome: Area Under the Plasma Drug Concentration Versus Time Curve (AUC[0-t]) Following Single Dose of GSK3145095 on Day 1-Part 1
Description: Blood samples were collected at the indicated time points for the determination of AUC(0-t) following single dose of GSK3145095 on Day 1 and was calculated by standard non-compartmental analysis.
Time Frame: Day 1:Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post-dose
Population: Pharmacokinetic (PK) Population. The PK Population consisted of all participants from the All-Treated Population for whom a PK sample was obtained and analyzed. Study was terminated in Part-1 during first escalation cohort "GSK3145095 50 mg BID", hence subsequent escalation cohorts were not initiated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanograms per milliliter
Arm/Group | Part 1-GSK3145095 50 mg BID | Part 1-GSK3145095 100 mg BID | Part 1-GSK3145095 200 mg BID | Part 1-GSK3145095 400 mg BID | Part 1-GSK3145095 800 mg BID
Number analyzed (Participants) | 8 | 0 | 0 | 0 | 0
Hour*nanograms per milliliter | 17411.6 (13.0) |  |  |  |

20. Secondary Outcome: AUC (0-t) Following Single Dose of GSK3145095 on Day 1-Part 2
Description: Blood samples were to be collected at the indicated time points for the determination of AUC (0-t) following single dose of GSK3145095 on Day 1 and was to be calculated by standard non-compartmental analysis.
Time Frame: Day 1:Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post-dose
Population: PK Population: Data were not collected for this endpoint as study was terminated during Part 1. Subsequent Part 2 was not initiated.
Arm/Group | Part 2-GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

21. Secondary Outcome: Area Under the Concentration-time Curve Over the Dosing Interval (AUC [0-tau]) Following Single Dose of GSK3145095 on Day 1-Part 1
Description: Blood samples were collected at the indicated time points for the determination of AUC (0-tau) following single dose of GSK3145095 on Day 1 and was calculated by standard non-compartmental analysis.
Time Frame: Day 1:Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post-dose
Population: PK Population: Study was terminated in Part-1 during first escalation cohort "GSK3145095 50 mg BID", hence subsequent escalation cohorts were not initiated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanograms per milliliter
Arm/Group | Part 1-GSK3145095 50 mg BID | Part 1-GSK3145095 100 mg BID | Part 1-GSK3145095 200 mg BID | Part 1-GSK3145095 400 mg BID | Part 1-GSK3145095 800 mg BID
Number analyzed (Participants) | 8 | 0 | 0 | 0 | 0
Hour*nanograms per milliliter | 11263.4 (19.2) |  |  |  |

22. Secondary Outcome: AUC (0-tau) Following Single Dose of GSK3145095 on Day 1-Part 2
Description: Blood samples were to be collected at the indicated time points for the determination of AUC (0-tau) following single dose of GSK3145095.
Time Frame: Day 1:Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post-dose
Population: as for outcome 20
Arm/Group | Part 2-GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

23. Secondary Outcome: Maximum Observed Plasma Drug Concentration (Cmax) Following Single Dose of GSK3145095 on Day 1-Part 1
Description: Blood samples were collected at the indicated time points for the determination of Cmax following single dose of GSK3145095 on Day 1 and was calculated by standard non-compartmental analysis.
Time Frame: Day 1:Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post-dose
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part 1-GSK3145095 50 mg BID | Part 1-GSK3145095 100 mg BID | Part 1-GSK3145095 200 mg BID | Part 1-GSK3145095 400 mg BID | Part 1-GSK3145095 800 mg BID
Number analyzed (Participants) | 8 | 0 | 0 | 0 | 0
Nanograms per milliliter | 1435.0 (25.7) |  |  |  |

24. Secondary Outcome: Cmax Following Single Dose of GSK3145095 on Day 1-Part 2
Description: Blood samples were to be collected at the indicated time points for the determination of Cmax following single dose of GSK3145095 on Day 1.
Time Frame: Day 1:Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post-dose
Population: as for outcome 20
Arm/Group | Part 2-GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

25. Secondary Outcome: Minimum Observed Plasma Drug Concentration (Cmin) Following Single Dose of GSK3145095 on Day 1-Part 1
Description: Blood samples were collected at the indicated time points for the determination of Cmin following single dose of GSK3145095 on Day 1 and was calculated by standard non-compartmental analysis.
Time Frame: Day 1:Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post-dose
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part 1-GSK3145095 50 mg BID | Part 1-GSK3145095 100 mg BID | Part 1-GSK3145095 200 mg BID | Part 1-GSK3145095 400 mg BID | Part 1-GSK3145095 800 mg BID
Number analyzed (Participants) | 8 | 0 | 0 | 0 | 0
Nanograms per milliliter | 344.8 (20.0) |  |  |  |

26. Secondary Outcome: Cmin Following Single Dose of GSK3145095 on Day 1-Part 2
Description: Blood samples were to be collected at the indicated time points for the determination of Cmin following single dose of GSK3145095 on Day 1.
Time Frame: Day 1:Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post-dose
Population: as for outcome 20
Arm/Group | Part 2-GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

27. Secondary Outcome: Time to Maximum Observed Plasma Drug Concentration (Tmax) Following Single Dose of GSK3145095 on Day 1-Part 1
Description: Blood samples were collected at the indicated time points for the determination of tmax following single dose of GSK3145095 on Day 1 and was calculated by standard non-compartmental analysis.
Time Frame: Day 1:Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post-dose
Population: as for outcome 21
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1-GSK3145095 50 mg BID | Part 1-GSK3145095 100 mg BID | Part 1-GSK3145095 200 mg BID | Part 1-GSK3145095 400 mg BID | Part 1-GSK3145095 800 mg BID
Number analyzed (Participants) | 8 | 0 | 0 | 0 | 0
Hours | 2.100 [1.57 to 5.83] |  |  |  |

28. Secondary Outcome: Tmax Following Single Dose of GSK3145095 on Day 1-Part 2
Description: Blood samples were to be collected at the indicated time points for the determination of tmax following single dose of GSK3145095 on Day 1.
Time Frame: Day 1:Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post-dose
Population: as for outcome 20
Arm/Group | Part 2-GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

29. Secondary Outcome: Clearance (CL/F) Following Single Dose of GSK3145095 on Day 1-Part 1
Description: Blood samples were collected at the indicated time points for the determination of CL/F following single dose of GSK3145095 on Day 1 and was calculated by standard non-compartmental analysis.
Time Frame: Day 1:Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post-dose
Population: PK Population: Only those participants with data available at the specified data points were analyzed. Study was terminated in Part-1 during first escalation cohort "GSK3145095 50 mg BID", hence subsequent escalation cohorts were not initiated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Groups:
- 1-GSK3145095 200 mg BID: Participants were to receive a single 400 mg dose of GSK3145095 orally on Day 1. From study Day 2, participants were to receive 800 mg dose of GSK3145095 given as 400 mg BID.
Arm/Group | Part 1-GSK3145095 50 mg BID | Part 1-GSK3145095 100 mg BID | Part 1-GSK3145095 200 mg BID | 1-GSK3145095 200 mg BID | Part 1-GSK3145095 800 mg BID
Number analyzed (Participants) | 6 | 0 | 0 | 0 | 0
Liters per hour | 2.149 (10.9) |  |  |  |

30. Secondary Outcome: CL/F Following Single Dose of GSK3145095 on Day 1-Part 2
Description: Blood samples were to be collected at the indicated time points for the determination of CL/F following single dose of GSK3145095 on Day 1.
Time Frame: Day 1:Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post-dose
Population: as for outcome 20
Arm/Group | Part 2-GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

31. Secondary Outcome: Volume of Distribution (Vz/F) Following Single Dose of GSK3145095 on Day 1-Part 1
Description: Blood samples were collected at the indicated time points for the determination of Vz/F following single dose of GSK3145095 on Day 1 and was calculated by standard non-compartmental analysis.
Time Frame: Day 1:Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post-dose
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Part 1-GSK3145095 50 mg BID | Part 1-GSK3145095 100 mg BID | Part 1-GSK3145095 200 mg BID | Part 1-GSK3145095 400 mg BID | Part 1-GSK3145095 800 mg BID
Number analyzed (Participants) | 6 | 0 | 0 | 0 | 0
Liters | 32.89 (17.3) |  |  |  |

32. Secondary Outcome: Vz/F Following Single Dose of GSK3145095 on Day 1-Part 2
Description: Blood samples were to be collected at the indicated time points for the determination of V/F following single dose of GSK3145095 on Day 1.
Time Frame: Day 1:Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post-dose
Population: as for outcome 20
Arm/Group | Part 2-GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

33. Secondary Outcome: Terminal Half-life (t1/2) Following Single Dose of GSK3145095 on Day 1-Part 1
Description: Blood samples were collected at the indicated time points for the determination of t1/2 following single dose of GSK3145095 on Day 1 and was calculated by standard non-compartmental analysis.
Time Frame: Day 1:Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post-dose
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | Part 1-GSK3145095 50 mg BID | Part 1-GSK3145095 100 mg BID | Part 1-GSK3145095 200 mg BID | Part 1-GSK3145095 400 mg BID | Part 1-GSK3145095 800 mg BID
Number analyzed (Participants) | 6 | 0 | 0 | 0 | 0
Hour | 10.608 (14.1) |  |  |  |

34. Secondary Outcome: T1/2 Following Single Dose of GSK3145095 on Day 1-Part 2
Description: Blood samples were to be collected at the indicated time points for the determination of t1/2 following single dose of GSK3145095 on Day 1.
Time Frame: Day 1:Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post-dose
Population: as for outcome 20
Arm/Group | Part 2-GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

35. Secondary Outcome: AUC (0-t) Following Repeat Dose of GSK3145095 on Day 15-Part 1
Description: Blood samples were collected at the indicated time points for the determination of AUC (0-t) following repeat dose of GSK3145095 on Day 15 and was calculated by standard non-compartmental analysis.
Time Frame: Day 15: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post dose
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanograms per milliliter
Arm/Group | Part 1-GSK3145095 50 mg BID | Part 1-GSK3145095 100 mg BID | Part 1-GSK3145095 200 mg BID | Part 1-GSK3145095 400 mg BID | Part 1-GSK3145095 800 mg BID
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
Hour*nanograms per milliliter | 19110.5 (56.3) |  |  |  |

36. Secondary Outcome: AUC (0-t) Following Repeat Dose of GSK3145095 on Day 15-Part 2
Description: Blood samples were to be collected at the indicated time points for the determination of AUC (0-t) following repeat dose of GSK3145095 on Day 15.
Time Frame: Day 15:Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post-dose
Population: as for outcome 20
Arm/Group | Part 2-GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

37. Secondary Outcome: AUC (0-tau) Following Repeat Dose of GSK3145095 on Day 15-Part 1
Description: Blood samples were collected at the indicated time points for the determination of AUC (0-tau) following repeat dose of GSK3145095 on Day 15 and was calculated by standard non-compartmental analysis.
Time Frame: Day 15: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post dose
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanograms per milliliter
Arm/Group | Part 1-GSK3145095 50 mg BID | Part 1-GSK3145095 100 mg BID | Part 1-GSK3145095 200 mg BID | Part 1-GSK3145095 400 mg BID | Part 1-GSK3145095 800 mg BID
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
Hour*nanograms per milliliter | 19110.5 (56.3) |  |  |  |

38. Secondary Outcome: AUC (0-tau) Following Repeat Dose of GSK3145095 on Day 15-Part 2
Description: Blood samples were to be collected at the indicated time points for the determination of AUC (0-tau) following repeat dose of GSK3145095 on Day 15.
Time Frame: Day 15:Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post-dose
Population: as for outcome 20
Arm/Group | Part 2-GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

39. Secondary Outcome: Cmax Following Repeat Dose of GSK3145095 on Day 15-Part 1
Description: Blood samples were collected at the indicated time points for the determination of Cmax following repeat dose of GSK3145095 on Day 15 and was calculated by standard non-compartmental analysis.
Time Frame: Day 15: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post dose
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part 1-GSK3145095 50 mg BID | Part 1-GSK3145095 100 mg BID | Part 1-GSK3145095 200 mg BID | Part 1-GSK3145095 400 mg BID | Part 1-GSK3145095 800 mg BID
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
Nanograms per milliliter | 2104.4 (42.0) |  |  |  |

40. Secondary Outcome: Cmax Following Repeat Dose of GSK3145095 on Day 15-Part 2
Description: Blood samples were to be collected at the indicated time points for the determination of Cmax following repeat dose of GSK3145095 on Day 15.
Time Frame: Day 15:Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post-dose
Population: as for outcome 20
Arm/Group | Part 2-GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

41. Secondary Outcome: Cmin Following Repeat Dose of GSK3145095 on Day 15-Part 1
Description: Blood samples were collected at the indicated time points for the determination of Cmin following repeat dose of GSK3145095 on day 15 and was calculated by standard non-compartmental analysis.
Time Frame: Day 15: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post dose
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part 1-GSK3145095 50 mg BID | Part 1-GSK3145095 100 mg BID | Part 1-GSK3145095 200 mg BID | Part 1-GSK3145095 400 mg BID | Part 1-GSK3145095 800 mg BID
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
Nanograms per milliliter | 953.6 (114.5) |  |  |  |

42. Secondary Outcome: Cmin Following Repeat Dose of GSK3145095 on Day 15-Part 2
Description: Blood samples were to be collected at the indicated time points for the determination of Cmin following repeat dose of GSK3145095 on Day 15.
Time Frame: Day 15:Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post-dose
Population: as for outcome 20
Arm/Group | Part 2-GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

43. Secondary Outcome: Tmax Following Repeat Dose of GSK3145095 on Day 15-Part 1
Description: Blood samples were collected at the indicated time points for the determination of tmax following repeat dose of GSK3145095 and was calculated by standard non-compartmental analysis.
Time Frame: Day 15: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post dose
Population: as for outcome 29
Measure: Median (Full Range); unit: Hour
Arm/Group | Part 1-GSK3145095 50 mg BID | Part 1-GSK3145095 100 mg BID | Part 1-GSK3145095 200 mg BID | Part 1-GSK3145095 400 mg BID | Part 1-GSK3145095 800 mg BID
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
Hour | 2.575 [2.12 to 7.97] |  |  |  |

44. Secondary Outcome: Tmax Following Repeat Dose of GSK3145095 on Day 15-Part 2
Description: Blood samples were to be collected at the indicated time points for the determination of tmax following repeat dose of GSK3145095 on Day 15.
Time Frame: Day 15:Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post-dose
Population: as for outcome 20
Arm/Group | Part 2-GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

45. Secondary Outcome: CL/F Following Repeat Dose of GSK3145095 on Day 15-Part 1
Description: Blood samples were collected at the indicated time points for the determination of CL/F following repeat dose of GSK3145095 on Day 15. For accurate estimation of CL/F following repeated administration, it is imperative that steady state has been achieved. As the attainment of steady state could not be confirmed with certainty, CL/F was not computed following repeated dose.
Time Frame: Day 15: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post dose
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Part 1-GSK3145095 50 mg BID | Part 1-GSK3145095 100 mg BID | Part 1-GSK3145095 200 mg BID | Part 1-GSK3145095 400 mg BID | Part 1-GSK3145095 800 mg BID
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
Liters per hour | NA (NA) — For accurate estimation of CL/F following repeated administration, it is imperative that steady state has been achieved. As the attainment of steady state could not be confirmed with certainty, CL/F was not computed following repeated dose. |  |  |  |

46. Secondary Outcome: CL/F Following Repeat Dose of GSK3145095 on Day 15-Part 2
Description: Blood samples were to be collected at the indicated time points for the determination of CL/F following repeat dose of GSK3145095 on Day 15.
Time Frame: Day 15:Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post-dose
Population: as for outcome 20
Arm/Group | Part 2-GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

47. Secondary Outcome: Vz/F Following Repeat Dose of GSK3145095 on Day 15-Part 1
Description: Blood samples were collected at the indicated time points for the determination of Vz/F following repeat dose of GSK3145095 on Day 15. As t1/2 following repeated administration could not be computed, Vz/F whose estimation is dependent upon the t1/2 could not be estimated as well.
Time Frame: Day 15: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post dose
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Part 1-GSK3145095 50 mg BID | Part 1-GSK3145095 100 mg BID | Part 1-GSK3145095 200 mg BID | Part 1-GSK3145095 400 mg BID | Part 1-GSK3145095 800 mg BID
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
Liters | NA (NA) — As t1/2 following repeated administration could not be computed, Vz/F whose estimation is dependent upon the t1/2 could not be estimated as well. |  |  |  |

48. Secondary Outcome: Vz/F Following Repeat Dose of GSK3145095 on Day 15-Part 2
Description: Blood samples were to be collected at the indicated time points for the determination of V/F following repeat dose of GSK3145095 on Day 15.
Time Frame: Day 15:Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post-dose
Population: as for outcome 20
Arm/Group | Part 2-GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

49. Secondary Outcome: T1/2 Following Repeat Dose of GSK3145095 on Day 15-Part 1
Description: Blood samples were collected at the indicated time points for the determination of t1/2 following repeat dose of GSK3145095 on Day 15. t1/2 following repeated administration was not computed because duration of observation (12 hours from the morning dose) was too short (less than 2 times the average half-life observed after the first dose) for its accurate estimation.
Time Frame: Day 15: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post dose
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | Part 1-GSK3145095 50 mg BID | Part 1-GSK3145095 100 mg BID | Part 1-GSK3145095 200 mg BID | Part 1-GSK3145095 400 mg BID | Part 1-GSK3145095 800 mg BID
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
Hour | NA (NA) — t1/2 following repeated administration was not computed because duration of observation (12 hours from the morning dose) was too short (less than 2 times the average half-life observed after the first dose) for its accurate estimation. |  |  |  |

50. Secondary Outcome: T1/2 Following Repeat Dose of GSK3145095 on Day 15-Part 2
Description: Blood samples were to be collected at the indicated time points for the determination of t1/2 following repeat dose of GSK3145095 on Day 15.
Time Frame: Day 15:Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post-dose
Population: as for outcome 20
Arm/Group | Part 2-GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

51. Secondary Outcome: Dose Proportionality of GSK3145095 for Dose Levels 100 mg (50 mg BID) to 1600 mg (800 mg BID) Using AUC (0-t) Following Single Dose-Part 1
Description: Dose proportionality was to be evaluated for GSK3145095 using a fixed effects power model. Estimated slope was to be presented to express dose proportionality. As only one dose level (100 mg) was tested prior to termination of the study and multiple dose levels are required to investigate dose proportionality, hence dose proportionality could not be analyzed.
Time Frame: Day 1: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post dose
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: Slope of log dose
Groups:
- Part 1-GSK3145095 50 mg BID to 800 mg BID: Participants in this arm received 100 mg as 50 mg BID dose of GSK3142095. From study Day 2 participants were to receive 200 mg as dose of 100 mg BID, 400 mg as dose of 200 mg BID, 800 mg as dose of 400 mg BID, 1600 mg as dose of 800 mg BID orally.
Arm/Group | Part 1-GSK3145095 50 mg BID to 800 mg BID
Number analyzed (Participants) | 8
Slope of log dose | NA [NA to NA] — As only one dose level (100 mg) was tested prior to termination of the study and multiple dose levels are required to investigate dose proportionality, hence dose proportionality could not be analyzed.

52. Secondary Outcome: Dose Proportionality of GSK3145095 for Dose Levels 100 mg (50 mg BID) to 1600 mg (800 mg) BID Using Cmax Following Single Dose-Part 1
Description: as for outcome 51
Time Frame: Day 1: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post dose
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: Slope of log dose
Arm/Group | Part 1-GSK3145095 50 mg BID to 800 mg BID
Number analyzed (Participants) | 8
Slope of log dose | NA [NA to NA] — As only one dose level (100 mg) was tested prior to termination of the study and multiple dose levels are required to investigate dose proportionality, hence dose proportionality could not be analyzed.

53. Secondary Outcome: Dose Proportionality of GSK3145095 for Dose Levels 100 mg (50 mg BID) to 1600 mg (800 mg BID) Using AUC (0-tau) Following Repeat Dose-Part 1
Description: as for outcome 51
Time Frame: Day 15: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post dose
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: Slope of log dose
Arm/Group | Part 1-GSK3145095 50 mg BID to 800 mg BID
Number analyzed (Participants) | 8
Slope of log dose | NA [NA to NA] — As only one dose level (100 mg) was tested prior to termination of the study and multiple dose levels are required to investigate dose proportionality, hence dose proportionality could not be analyzed.

54. Secondary Outcome: Dose Proportionality of GSK3145095 for Dose Levels 100 mg (50 mg BID) to 1600 mg (800 mg BID) Using Cmax Following Repeat Dose-Part 1
Description: as for outcome 51
Time Frame: Day 15: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post dose
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: Slope of log dose
Arm/Group | Part 1-GSK3145095 50 mg BID to 800 mg BID
Number analyzed (Participants) | 8
Slope of log dose | NA [NA to NA] — As only one dose level (100 mg) was tested prior to termination of the study and multiple dose levels are required to investigate dose proportionality, hence dose proportionality could not be analyzed.

55. Secondary Outcome: Dose Proportionality of GSK3145095 Using AUC (0-t) Following Single Dose-Part 2
Description: Dose proportionality was to be evaluated for GSK3145095 using a fixed effects power model. Estimated slope was to be presented to express dose proportionality.
Time Frame: Day 1: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post dose
Population: as for outcome 20
Arm/Group | Part 2- GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

56. Secondary Outcome: Dose Proportionality of GSK3145095 Using Cmax Following Single Dose-Part 2
Description: as for outcome 55
Time Frame: Day 1: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post dose
Population: as for outcome 20
Arm/Group | Part 2- GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

57. Secondary Outcome: Dose Proportionality of GSK3145095 Using AUC (0-tau) Following Repeat Dose-Part 2
Description: as for outcome 55
Time Frame: Day 15: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8,10, and 24 hours post dose
Population: as for outcome 20
Arm/Group | Part 2- GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

58. Secondary Outcome: Dose Proportionality Using Cmax Following Repeat Dose of GSK3145095-Part 2
Description: as for outcome 55
Time Frame: Day 15: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post dose
Population: as for outcome 20
Arm/Group | Part 2- GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

59. Secondary Outcome: Accumulation Ratio Following Repeat Dose of GSK3145095 on Day 15-Part 1
Description: Accumulation ratio was calculated as AUC(0-tau) at Day 15 divided by AUC(0-tau) at Day 1 for GSK3145095.
Time Frame: Day 1: Pre-dose,0.5,1,1.5,2,3,4,6,8, 10, and 24 hour post-dose, Days 15: Pre-dose,0.5,1,1.5,2,3,4,6,8,10,24 hour post dose
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of AUC
Arm/Group | Part 1-GSK3145095 50 mg BID | Part 1-GSK3145095 100 mg BID | Part 1-GSK3145095 200 mg BID | Part 1-GSK3145095 400 mg BID | Part 1-GSK3145095 800 mg BID
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
Ratio of AUC | 1.792 (57.5) |  |  |  |

60. Secondary Outcome: Accumulation Ratio Following Repeat Dose of GSK3145095 on Day 15-Part 2
Description: Accumulation ratio was to be calculated as AUC(0-tau) at Day 15 divided by AUC(0-tau) at Day 1 for GSK3145095.
Time Frame: as for outcome 59
Population: as for outcome 20
Arm/Group | Part 2-GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

61. Secondary Outcome: Time Invariance of GSK3145095-Part 1
Description: Blood samples were collected at indicated time points for analysis of time invariance. Time invariance was calculated as AUC(0-tau) at Day 15 divided by AUC(0-infinity) at Day 1 for GSK3145095.
Time Frame: Day 1: Pre-dose,0.5,1,1.5,2,3,4,6,8,10, and 24 hour post-dose, Days 15: Pre-dose,0.5,1,1.5,2,3,4,6,8,10,24 hour post dose
Population: as for outcome 29
Measure: Median (Full Range); unit: Ratio
Arm/Group | Part 1-GSK3145095 50 mg BID | Part 1-GSK3145095 100 mg BID | Part 1-GSK3145095 200 mg BID | Part 1-GSK3145095 400 mg BID | Part 1-GSK3145095 800 mg BID
Number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
Ratio | 0.78 [0.71 to 0.85] |  |  |  |

62. Secondary Outcome: Time Invariance of GSK3145095-Part 2
Description: Blood samples were to be collected at indicated time points for analysis of time invariance. Time invariance were to be calculated as AUC(0-tau) at Day 15 divided by AUC(0-infinity) at Day 1 for GSK3145095.
Time Frame: Day 1: Pre-dose,0.5,1,1.5,2,3,4,6,8, 10, and 24 hour post-dose, Days 15: Pre-dose,0.5,1,1.5,2,3,4,6,8,10, and 24 hour post dose
Population: as for outcome 20
Arm/Group | Part 2-GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

63. Secondary Outcome: Plasma Concentration of Pembrolizumab -Part 2
Description: Blood samples were to be collected at indicated time points for the determination of plasma concentration of pembrolizumab.
Time Frame: Day 1: pre-dose, 0.5 hour (within 30 minutes after end of infusion), 24 hours after end of infusion; Days 8,15 (anytime during visit); Days 22,43,64 and every 21 days thereafter (pre-dose), for up to 2 years
Population: as for outcome 20
Arm/Group | Part 2-GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

64. Secondary Outcome: Cmax of Pembrolizumab-Part 2
Description: Blood samples were to be collected at indicated time points for the determination of Cmax of pembrolizumab.
Time Frame: as for outcome 63
Population: as for outcome 20
Arm/Group | Part 2-GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

65. Secondary Outcome: AUC (0-tau) of Pembrolizumab-Part 2
Description: Blood samples were to be collected at indicated time points for the determination of AUC (0-tau) of pembrolizumab.
Time Frame: as for outcome 63
Population: as for outcome 20
Arm/Group | Part 2-GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

66. Secondary Outcome: Cmin of Pembrolizumab-Part 2
Description: Blood samples were to be collected at indicated time points for the determination of Cmin of pembrolizumab.
Time Frame: as for outcome 63
Population: as for outcome 20
Arm/Group | Part 2-GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

67. Secondary Outcome: AUC (0-t) Following Single Dose of GSK3145095 on Day 1-Part 3
Description: Blood samples were to be collected at the indicated time points for the determination of AUC (0-t) following single dose of GSK3145095 on Day 1.
Time Frame: Day 1:Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post-dose
Population: PK Population: Data were not collected for this endpoint as study was terminated during Part 1. Subsequent Part 3 was not initiated.
Arm/Group | Part 3 GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

68. Secondary Outcome: Cmax Following Single Dose of GSK3145095 on Day 1-Part 3
Description: as for outcome 24
Time Frame: Day 1:Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post-dose
Population: as for outcome 67
Arm/Group | Part 3 GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

69. Secondary Outcome: Tmax Following Single Dose of GSK3145095 on Day 1-Part 3
Description: as for outcome 28
Time Frame: Day 1:Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post-dose
Population: as for outcome 67
Arm/Group | Part 3 GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

70. Secondary Outcome: T1/2 Following Single Dose of GSK3145095 on Day 1-Part 3
Description: as for outcome 34
Time Frame: Day 1:Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post-dose
Population: as for outcome 67
Arm/Group | Part 3 GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

71. Secondary Outcome: AUC (0-t) Following Repeat Dose of GSK3145095 on Day 15-Part 3
Description: as for outcome 36
Time Frame: Day 15:Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 hours post-dose
Population: as for outcome 67
Arm/Group | Part 3 GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

72. Secondary Outcome: Cmax Following Repeat Dose of GSK3145095 on Day 15-Part 3
Description: as for outcome 40
Time Frame: Day 15:Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 hours post-dose
Population: as for outcome 67
Arm/Group | Part 3 GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

73. Secondary Outcome: Tmax Following Repeat Dose of GSK3145095 on Day 15-Part 3
Description: as for outcome 44
Time Frame: Day 15:Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 hours post-dose
Population: as for outcome 67
Arm/Group | Part 3 GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

74. Secondary Outcome: T1/2 Following Repeat Dose of GSK3145095 on Day 15-Part 3
Description: as for outcome 50
Time Frame: Day 15:Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 hours post-dose
Population: as for outcome 67
Arm/Group | Part 3 GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

75. Secondary Outcome: AUC (0-t) Following Single Dose of Pembrolizumab-Part 3
Description: Blood samples were to be collected at the indicated time points for the determination of AUC (0-t) following single dose of pembrolizumab.
Time Frame: Day 1: pre-dose, 0.5 hour (within 30 minutes after end of infusion), 24 hour after end of infusion
Population: as for outcome 67
Arm/Group | Part 3 GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

76. Secondary Outcome: AUC (0-tau) Following Single Dose of Pembrolizumab -Part 3
Description: Blood samples were to be collected at the indicated time points for the determination of AUC (0-tau) following single dose of pembrolizumab.
Time Frame: Day 1: pre-dose, 0.5 hour (within 30 minutes after end of infusion), 24 hour after end of infusion
Population: as for outcome 67
Arm/Group | Part 3 GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

77. Secondary Outcome: Cmax Following Single Dose of Pembrolizumab -Part 3
Description: Blood samples were to be collected at the indicated time points for the determination of Cmax following single dose of pembrolizumab.
Time Frame: Day 1: pre-dose, 0.5 hour (within 30 minutes after end of infusion), 24 hour after end of infusion
Population: as for outcome 67
Arm/Group | Part 3 GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

78. Secondary Outcome: Tmax Following Single Dose of Pembrolizumab -Part 3
Description: Blood samples were to be collected at the indicated time points for the determination of tmax following single dose of pembrolizumab.
Time Frame: Day 1: pre-dose, 0.5 hour (within 30 minutes after end of infusion), 24 hour after end of infusion
Population: as for outcome 67
Arm/Group | Part 3 GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

79. Secondary Outcome: T1/2 Following Single Dose of Pembrolizumab -Part 3
Description: Blood samples were to be collected at the indicated time points for the determination of t1/2 following single dose of pembrolizumab.
Time Frame: Day 1: pre-dose, 0.5 hour (within 30 minutes after end of infusion), 24 hour after end of infusion
Population: as for outcome 67
Arm/Group | Part 3 GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

80. Secondary Outcome: AUC (0-t) Following Repeat Dose of Pembrolizumab -Part 3
Description: Blood samples were to be collected at the indicated time points for the determination of AUC (0-t) following repeat dose of pembrolizumab.
Time Frame: as for outcome 63
Population: as for outcome 67
Arm/Group | Part 3 GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

81. Secondary Outcome: AUC (0-tau) Following Repeat Dose of Pembrolizumab -Part 3
Description: Blood samples were to be collected at the indicated time points for the determination of AUC (0-tau) following repeat dose of pembrolizumab.
Time Frame: as for outcome 63
Population: as for outcome 67
Arm/Group | Part 3 GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

82. Secondary Outcome: Cmax Following Repeat Dose of Pembrolizumab -Part 3
Description: Blood samples were to be collected at the indicated time points for the determination of Cmax following repeat dose of pembrolizumab.
Time Frame: as for outcome 63
Population: as for outcome 67
Arm/Group | Part 3 GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

83. Secondary Outcome: Tmax Following Repeat Dose of Pembrolizumab -Part 3
Description: Blood samples were to be collected at the indicated time points for the determination of tmax following repeat dose of pembrolizumab.
Time Frame: as for outcome 63
Population: as for outcome 67
Arm/Group | Part 3 GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

84. Secondary Outcome: T1/2 Following Repeat Dose of Pembrolizumab -Part 3
Description: Blood samples were to be collected at the indicated time points for the determination of t1/2 following repeat dose of pembrolizumab.
Time Frame: as for outcome 63
Population: as for outcome 67
Arm/Group | Part 3 GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

85. Secondary Outcome: Dose Proportionality of GSK3145095 Using AUC (0-t) Following Single Dose-Part 3
Description: as for outcome 55
Time Frame: Day 1:Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post-dose
Population: as for outcome 67
Arm/Group | Part 3 GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

86. Secondary Outcome: Dose Proportionality of GSK3145095 Using Cmax Following Single Dose-Part 3
Description: as for outcome 55
Time Frame: Day 1:Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post-dose
Population: as for outcome 67
Arm/Group | Part 3 GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

87. Secondary Outcome: Dose Proportionality of GSK3145095 Using AUC (0-tau) Following Repeat Dose of GSK3145095-Part 3
Description: as for outcome 55
Time Frame: Day 15: Pre-dose,0.5,1,1.5,2,3,4,6,8,10,24 hour post morning dose; Day 15: 0.5,1,2,3,6,8 hour post evening dose
Population: as for outcome 67
Arm/Group | Part 3 GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

88. Secondary Outcome: Dose Proportionality of GSK3145095 Using Cmax Following Repeat Dose-Part 3
Description: as for outcome 55
Time Frame: Day 15: Pre-dose,0.5,1,1.5,2,3,4,6,8,10,24 hour post morning dose; Day 15: 0.5,1,2,3,6,8 hour post evening dose
Population: as for outcome 67
Arm/Group | Part 3 GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

89. Secondary Outcome: Accumulation Ratio Following Repeat Dose of GSK3145095-Part 3
Description: Accumulation ratio was to be calculated as AUC(0-tau) at Day 15 divided by AUC(0-tau) at Day 1 for GSK3145095.
Time Frame: Days 1: Pre-dose,0.5,1,1.5,2,3,4,6,8,10,24 hour post-dose; Day 15: Pre-dose,0.5,1,1.5,2,3,4,6,8,10,24 hour post morning dose; Day 15: 0.5,1,2,3,6,8 hour post evening dose
Population: as for outcome 67
Arm/Group | Part 3 GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

90. Secondary Outcome: Time Invariance Following Repeat Dose of GSK3145095-Part 3
Description: Blood samples were to be collected at indicated time points for analysis of time invariance. Time invariance was to be calculated as AUC(0-tau) at Day 15 divided by AUC(0-infinity) at Day 1 for GSK3145095.
Time Frame: Days 1: Pre - dose ,0.5,1,1.5,2,3,4,6,8,10,24 hour; Day 15: Pre - dose ,0.5,1,1.5,2,3,4,6,8,10,24 hour post morning dose ; Day 15:0.5,1,2,3,6,8 hour post evening dose
Population: as for outcome 67
Arm/Group | Part 3 GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

91. Secondary Outcome: Dose Proportionality for Pembrolizumab Using AUC (0-t) Following Single Dose-Part 3
Description: as for outcome 55
Time Frame: Day 1: pre-dose, 0.5 hour (within 30 minutes after end of infusion), 24 hour after end of infusion
Population: as for outcome 67
Arm/Group | Part 3 GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

92. Secondary Outcome: Dose Proportionality for Pembrolizumab Using Cmax Following Single Dose-Part 3
Description: as for outcome 55
Time Frame: Day 1: pre-dose, 0.5 hour (within 30 minutes after end of infusion), 24 hour after end of infusion
Population: as for outcome 67
Arm/Group | Part 3 GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

93. Secondary Outcome: Dose Proportionality for Pembrolizumab Using AUC (0-tau) Following Repeat Dose-Part 3
Description: as for outcome 55
Time Frame: as for outcome 63
Population: as for outcome 67
Arm/Group | Part 3 GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

94. Secondary Outcome: Dose Proportionality for Pembrolizumab Using Cmax Following Repeat Dose-Part 3
Description: as for outcome 55
Time Frame: as for outcome 63
Population: as for outcome 67
Arm/Group | Part 3 GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

95. Secondary Outcome: Accumulation Ratio Following Repeat Dose of Pembrolizumab-Part 3
Description: Accumulation ratio was to be calculated as AUC(0-tau) at Day 15 divided by AUC(0-tau) at Day 1 for pembrolizumab.
Time Frame: Day 1: pre-dose, 0.5 hour (within 30 minutes after end of infusion), 24 hours after end of infusion; Day 15 (anytime during visit)
Population: as for outcome 67
Arm/Group | Part 3 GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

96. Secondary Outcome: Time Invariance Following Repeat Dose of Pembrolizumab-Part 3
Description: Blood samples were to be collected at indicated timepoints for analysis of time invariance. Time invariance was to be calculated as AUC(0-tau) at Day 15 divided by AUC(0-infinity) at Day 1 for pembrolizumab.
Time Frame: as for outcome 95
Population: as for outcome 67
Arm/Group | Part 3 GSK3145095+ Pembrolizumab 200 mg
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Non-serious AEs and SAEs were collected up to Day 95 in Part 1
Description: Non-serious AEs and SAEs were reported for all treated Population. Data is presented for Part 1 "GSK3145095 50 mg BID" only, as study was terminated during this first escalation cohort, hence subsequent escalation cohorts of Part-1 were not initiated. Parts 2, 3 and 4 were also not initiated.
Arm/Group | Part 1-GSK3145095 50 mg BID | Part 1-GSK3145095 100 mg BID | Part 1-GSK3145095 200 mg BID | Part 1-GSK3145095 400 mg BID | Part 1-GSK3145095 800 mg BID
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 4/8 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 8/8 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1-GSK3145095 50 mg BID (N=8) | Part 1-GSK3145095 100 mg BID (N=0) | Part 1-GSK3145095 200 mg BID (N=0) | Part 1-GSK3145095 400 mg BID (N=0) | Part 1-GSK3145095 800 mg BID (N=0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA | NA | NA | NA
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | NA | NA | NA | NA
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | NA | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 2 (2) | NA | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 1 (1) | NA | NA | NA | NA
Nausea (Gastrointestinal disorders) | 1 (1) | NA | NA | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1-GSK3145095 50 mg BID (N=8) | Part 1-GSK3145095 100 mg BID (N=0) | Part 1-GSK3145095 200 mg BID (N=0) | Part 1-GSK3145095 400 mg BID (N=0) | Part 1-GSK3145095 800 mg BID (N=0)
Constipation (Gastrointestinal disorders) | 3 (5) | NA | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 3 (3) | NA | NA | NA | NA
Abdominal distension (Gastrointestinal disorders) | 2 (3) | NA | NA | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 2 (5) | NA | NA | NA | NA
Nausea (Gastrointestinal disorders) | 2 (3) | NA | NA | NA | NA
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | NA | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 1 (1) | NA | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 1 (1) | NA | NA | NA | NA
Dyspepsia (Gastrointestinal disorders) | 1 (2) | NA | NA | NA | NA
Eructation (Gastrointestinal disorders) | 1 (1) | NA | NA | NA | NA
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | NA | NA | NA | NA
Lip swelling (Gastrointestinal disorders) | 1 (1) | NA | NA | NA | NA
Aspartate aminotransferase increased (Investigations) | 5 (7) | NA | NA | NA | NA
Alanine aminotransferase increased (Investigations) | 3 (4) | NA | NA | NA | NA
Blood alkaline phosphatase increased (Investigations) | 2 (4) | NA | NA | NA | NA
Lymphocyte count decreased (Investigations) | 2 (5) | NA | NA | NA | NA
Platelet count decreased (Investigations) | 2 (2) | NA | NA | NA | NA
Blood bilirubin increased (Investigations) | 1 (1) | NA | NA | NA | NA
Blood creatinine increased (Investigations) | 1 (1) | NA | NA | NA | NA
Weight decreased (Investigations) | 1 (1) | NA | NA | NA | NA
White blood cell count decreased (Investigations) | 1 (1) | NA | NA | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | NA | NA | NA | NA
Dehydration (Metabolism and nutrition disorders) | 1 (3) | NA | NA | NA | NA
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | NA | NA | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 4 (7) | NA | NA | NA | NA
Fatigue (General disorders) | 5 (7) | NA | NA | NA | NA
Anaemia (Blood and lymphatic system disorders) | 4 (6) | NA | NA | NA | NA
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | NA | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | NA | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | NA | NA | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | NA | NA | NA | NA
Clostridium difficile infection (Infections and infestations) | 1 (1) | NA | NA | NA | NA
Herpes zoster (Infections and infestations) | 1 (1) | NA | NA | NA | NA
Urinary tract infection (Infections and infestations) | 1 (1) | NA | NA | NA | NA
Dysgeusia (Nervous system disorders) | 1 (1) | NA | NA | NA | NA
Headache (Nervous system disorders) | 1 (1) | NA | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA | NA | NA | NA
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA | NA | NA | NA
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA | NA | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | NA | NA | NA | NA
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | NA | NA | NA | NA
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | NA | NA | NA | NA
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (3) | NA | NA | NA | NA
Jaundice (Hepatobiliary disorders) | 1 (1) | NA | NA | NA | NA
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | NA | NA | NA | NA
Anxiety (Psychiatric disorders) | 1 (1) | NA | NA | NA | NA
Depression (Psychiatric disorders) | 1 (1) | NA | NA | NA | NA
Insomnia (Psychiatric disorders) | 1 (1) | NA | NA | NA | NA
Chromaturia (Renal and urinary disorders) | 1 (1) | NA | NA | NA | NA
Renal failure (Renal and urinary disorders) | 1 (1) | NA | NA | NA | NA
Vaginal discharge (Reproductive system and breast disorders) | 1 (2) | NA | NA | NA | NA
Hypertension (Vascular disorders) | 1 (4) | NA | NA | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial

DOCUMENTS (2):
  • Study Protocol (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/51/NCT03681951/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-18): https://cdn.clinicaltrials.gov/large-docs/51/NCT03681951/SAP_001.pdf